CLINICAL TRIAL: NCT02898870
Title: Study of the Role of Occupational Exposure to Pesticides in the Prognosis of Lymphomas Diffuse Large B Cell in
Brief Title: Occupational Exposure to Pesticides in the Prognosis of Lymphomas
Acronym: ProLyPhy
Status: Terminated | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9668
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2016-09

CONDITIONS: Lymphoma Diffuse Large B-cell
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The link between the products of synthetic chemistry and cancer is at the heart of much research. Recent work has identified the use of plant protection agents by farmers as a risk factor for developing non-Hodgkin lymphoma, including diffuse large B cell lymphoma (DLBCL) is the most common histology. Different biological models were used to understand the role of pesticides in lymphomagenesis. To summarize, most pesticides act at the cellular and molecular level, on different signaling pathways. After metabolized by cytochrome P450, these compounds generally become pro-oxidants. The increase in reactive oxygen species rate (SAR) causes the activation of signaling pathways involved in cell proliferation and survival. But deregulation of oxidative status does not in itself justify the specificity of the impact of pesticides on specific pathologies. Several agents have a genotoxic effect, others induce the activation of signaling pathways by binding to transcription factors and others have immunomodulating properties.

DETAILED DESCRIPTION:
The link between the products of synthetic chemistry and cancer is at the heart of much research. Recent work has identified the use of plant protection agents by farmers as a risk factor for developing non-Hodgkin lymphoma, including diffuse large B cell lymphoma (DLBCL) is the most common histology. Different biological models were used to understand the role of pesticides in lymphomagenesis. To summarize, most pesticides act at the cellular and molecular level, on different signaling pathways. After metabolized by cytochrome P450, these compounds generally become pro-oxidants. The increase in reactive oxygen species rate (SAR) causes the activation of signaling pathways involved in cell proliferation and survival. But deregulation of oxidative status does not in itself justify the specificity of the impact of pesticides on specific pathologies. Several agents have a genotoxic effect, others induce the activation of signaling pathways by binding to transcription factors and others have immunomodulating properties.

Among these four mechanisms by which pesticides are involved in lymphomagenesis, two are also associated with resistance to chemotherapy. Thus, genotoxic agents leads the implementation process of DNA repair, used to repair genotoxic lesions induced by chemotherapeutic agents and evade apoptosis. On the other hand, to survive a high level of ROS, the tumor cell raises the level of antioxidant defenses, maintaining redox homeostasis and preventing oxidative stress. However, a high production of antioxidants constitutes a barrier to the effectiveness of anti-tumor agents which are effective in the generation of oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

Adults treated for diffuse large B-cell lymphoma:

* Diagnosed between 2010 and 2015
* Having received immuno-chemotherapy R-CHOP
* Supported in the health facilities of the Languedoc-Rousillon

Exclusion Criteria:

NA

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults treated for diffuse large B-cell lymphoma:
Sampling Method: Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2015-07; Primary Completion 2017-10 (Actual); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
pesticide exposure | 1 day
  The exposure measurement will be carried out using a self-administered questionnaire sent to patients on their professional activities. If farming a second questionnaire will further characterize the exposure to pesticides

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain LAMURE, Principal Investigator — University Hospital, Montpellier
Locations (1):
- LAMURE, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided